CLINICAL TRIAL: NCT02116075
Title: Caudal Corticosteroid vs. Dextrose Injection for Lumbosacral Radicular Pain.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Naveed Natanzi (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Naveed Natanzi, Resident Physician, VA Long Beach Healthcare System
Organization: VA Long Beach Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SC2626
Record Dates: First submitted 2014-04-09; First posted 2014-04-16 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: no Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Epidural Steroid (Experimental): 80mg depo-medrol 9mL 1% lidocaine
  Interventions: Procedure: Epidural Prolotherapy
- Epidural Prolotherapy (Active Comparator): 10ml of 5% generic dextrose
  Interventions: Procedure: Epidural Steroid

INTERVENTIONS:
Procedure: Epidural Prolotherapy — caudal injection of 10mL 5% dextrose
  Arms: Epidural Steroid
Procedure: Epidural Steroid — caudal injection of 1mL 80mg depo-medrol with 9ml of 1% lidocaine
  Arms: Epidural Prolotherapy

SUMMARY:
Study comparing caudal prolotherapy to conventional steroid for chronic low back pain

ELIGIBILITY:
INCLUSION CRITERIA

1. Participants must satisfy diagnostic criteria for lumbar radicular pain at L4 nerve root level or below with consistent MRI or X ray findings.
2. Evidence of low back pain base upon one or more of the following:

   i. Lumbar back pain episodes lasting greater than 6 months and current pain level is greater than 6/10 on VAS.

   ii. Has received at lest 2 types of ancillary treatment (i.e. physical therapy, oral analgesia, acupuncture, etc.)
3. Men or women age greater than or equal to 18 years.
4. No significant alcohol use (7 or fewer drinks per week).
5. Patient has a history of at least 2 failed epidural CS injections.

EXCLUSION CRITERIA

1. Treatment risk factors including one or more of the following:

   i. Unstable or symptomatic cardiac complaints ii. Unstable or symptomatic respiratory complaints iii. Unable to reliably comprehend the protocol or reliably record data
2. Pregnancy. A serum pregnancy test must be performed and negative in all women of child bearing potential within 2 weeks prior to enrollment.
3. History of Malignancy
4. Any medical (i.e. malignancy, infection, thrombo-embolic states, autoimmune disease, polyneuropathy) or psychosocial condition that in the opinion of the investigator, could jeopardize the subject's participation, and compliance with the study criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Pain relief as measured by VAS pain scale. | 1 year

SECONDARY OUTCOMES:
Change in the frequency and amount of opioid use. | 1 year
Disability score as determined by Oswstery questionnaire. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Veteran'S Affairs Healthy System, Long Beach, California, United States